CLINICAL TRIAL: NCT01326312
Title: Phase II, Open Label, Dose Finding Study of the Effect of GTx-758 on Total and Free Testosterone Levels in Men With Prostate Cancer Compared to a Luteinizing Hormone Releasing Hormone Agonist
Brief Title: Effect of GTx-758 on Total and Free Testosterone Levels in Men With Prostate Cancer
Acronym: GTx758
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: FDA Clinical Hold
Sponsor: GTx (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: G200705
Record Dates: First submitted 2011-03-25; First posted 2011-03-30 (Estimated); Results first posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2021-02

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — 3-fluoro-N-(4-fluorophenyl)-4-hydroxy-N-(4-hydroxyphenyl)benzamide; Leuprolide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- GTx- 758 1000mg (Experimental): GTx-758/Experimental/ nonsteroidal selective ER alpha agonist
  Interventions: Drug: GTx-758 2000mg
- GTx-758 2000mg (Experimental): GTx-758/Experimental/ nonsteroidal selective ER alpha agonist
  Interventions: Drug: GTx-758 1000mg
- Lupron Depot (Active Comparator): Luteinizing Hormone Releasing Hormone Agonist
  Interventions: Drug: Lupron Depot

INTERVENTIONS:
Drug: GTx-758 1000mg — comparison of different dosages of GTx-758 with leuprolide acetate for depot suspension
  Arms: GTx-758 2000mg
Drug: Lupron Depot — comparison of different dosages of GTx-758 with leuprolide acetate for depot suspension
  Arms: Lupron Depot
Drug: GTx-758 2000mg — comparison of different dosages of GTx-758 with leuprolide acetate for depot suspension
  Arms: GTx- 758 1000mg

SUMMARY:
The purpose of this study is to determine whether GTx 758 is effective in achieving and maintaining castrate testosterone levels in men with advanced prostate cancer.

DETAILED DESCRIPTION:
Prostate cancer is one of the most frequently diagnosed noncutaneous cancers among men in the US and is the second most common cause of cancer deaths. Patients with advanced prostate cancer undergo androgen deprivation therapy (ADT), by either LHRH agonists, LHRH antagonists, DES and other nonselective estrogens, or by bilateral orchiectomy. ADT by LHRH agonists, LHRH antagonists, or bilateral orchiectomy not only reduces testosterone, but also substantially lowers estrogen levels as estrogen is derived from the aromatization of testosterone. ADT-induced estrogen deficiency causes significant side effects which include hot flushes, gynecomastia, bone loss, decreases in bone quality and strength, osteoporosis and life-threatening fractures, adverse lipid changes, increase in body fat composition, and higher cardiovascular disease and myocardial infarction, and depression and other mood changes.

GTx-758 is a nonsteroidal selective ER agonist that suppresses LH secretion by the pituitary by feedback inhibition of the hypothalamic-pituitary-gonadal axis to induce castrate levels of testosterone. However, because it is a selective ER agonist, GTx-758 may maintain bone, does not induce hot flushes, avoids adverse lipid changes and body fat composition changes, and does not have the acute testosterone surge that are associated with other forms of ADT.

ELIGIBILITY:
Inclusion Criteria:

1. be between age 45 and 80 years of age
2. be able to communicate effectively with study personnel
3. ECOG is < or = 2
4. screening serum total testosterone> or = 150ng/dL
5. have prostate cancer, confirmed by pathology report
6. have not been treated with androgen deprivation therapy(chemical or surgical
7. have a clinical indication for the initiation of androgen deprivation therapy
8. give written informed consent prior to any study specific procedures
9. subject must agree to use acceptable methods of contraception

Exclusion Criteria:

1. known hypersensitivity or allergy to estrogen or estrogen like drugs
2. a clinically significant concurrent illness or psychological, familial, sociological, geographical or other concomitant condition that would not permit adequate follow-up and compliance with the study protocol
3. history of abnormal blood clotting,Factor V Leiden clotting disorder, thrombotic disease
4. have ALT or AST above 2 times the upper normal limit
5. have alkaline phosphatase greater than 3 times UNL and/or bilirubin levels above 2mg/dL at baseline
6. patients cannot have brain or spinal cord metastases
7. patients cannot have or be at risk for spinal cord compression from bone metastases
8. received an investigational drug within a period of 90 days prior to enrollment in the study
9. received the study medication previously
10. currently taking testosterone, testosterone-like agents, or antiandrogens including 5-alpha reductase inhibitors within 4 weeks of randomization
11. currently taking Saw Palmetto or PC-SPES (the subject may be considered for randomization after a 4 week washout period prior to randomization)
12. have taken diethylstilbestrol or other estrogen products within the previous 12 months prior to randomization
13. have taken body building or fertility supplements within 4 weeks of admission into the study (steroids and steroid like supplements)
14. have a history of cancer other than prostate cancer, superficial bladder cancer (with no recurrence in the last 5 years) and/or non-melanoma carcinoma of the skin
15. QTcB>480 msec, If the first QTcB reading exceeds 480msec two additional ECGs are to be performed separated at least 5 min apart, then take the average of the three QTcB or readings to determine if the subject satisfies the above criteria. If the average QYcB reading is >480 msec then the subject is excluded.

Ages: 45 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2011-06; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Steiner, MD, Study Director — GTx
Locations (36):
- United States (36):
  - GTx Investigative Site, Phoenix, Arizona
  - GTx Investigative Site, La Mesa, California
  - GTx Investigative Site, Los Angeles, California
  - GTx Investigative Site, San Bernardino, California
  - GTx Investigative Site, Middlebury, Connecticut
  - GTx Investigative Site, Aventura, Florida
  - GTx Investigative Site, Daytona Beach, Florida
  - GTx Investigative Site, Wellington, Florida
  - GTx Investigative Site, Marietta, Georgia
  - GTx Investigative Site, Springfield, Illinois
  - GTx Investigative Site, Fort Wayne, Indiana
  - GTx Investigative Site, Indianapolis, Indiana
  - GTx Investigative Site, Jeffersonville, Indiana
  - GTx Investigative Site, Annapolis, Maryland
  - GTx Investigative Site, Baltimore, Maryland
  - GTx Investigative Site, Brick, New Jersey
  - GTx Investigative Site, Lawrenceville, New Jersey
  - GTx Investigative Site, Albuquerque, New Mexico
  - GTx Investigative Site, Albany, New York
  - GTx Investigative Site, Garden City, New York
  - GTx Investigative Site, New York, New York
  - GTx Investigative Site, Oneida, New York
  - GTx Investigative Site, Syracuse, New York
  - GTx Investigative Site, Chapel Hill, North Carolina
  - GTx Investigative Site, Raleigh, North Carolina
  - GTx Investigative Site, Cincinnati, Ohio
  - GTx Investigative Site, Columbus, Ohio
  - GTx Investigative Site, Bala-Cynwyd, Pennsylvania
  - GTx Investigative Site, Lancaster, Pennsylvania
  - GTx Investigative Site, Pittsburgh, Pennsylvania
  - GTx Investigative Site, Myrtle Beach, South Carolina
  - GTx Investigative Site, Memphis, Tennessee
  - GTx Investigative Site, Nashville, Tennessee
  - GTx Investigative Site, Arlington, Texas
  - GTx Investigative Site, Houston, Texas
  - GTx Investigative Site, San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- GTx 758 1000mg; GTx-758 2000mg: GTx-758/Experimental/ nonsteroidal selective ER alpha agonist
  GTx-758: comparison of different dosages of GTx-758 with leuprolide acetate for depot suspension
Period: Overall Study
Arm/Group | GTx 758 1000mg | GTx-758 2000mg | Lupron Depot
Started | 53 | 55 | 51
Completed | 0 | 0 | 0
Not Completed | 53 | 55 | 51
Not completed — Adverse Event | 11 | 11 | 1
Not completed — Withdrawal by Subject | 1 | 2 | 1
Not completed — Protocol Violation | 0 | 1 | 0
Not completed — Lack of Efficacy | 13 | 7 | 1
Not completed — Death | 1 | 0 | 1
Not completed — progressive disease | 0 | 1 | 1
Not completed — Study terminated by Sponsor | 8 | 32 | 46
Not completed — Treatment arm terminated | 19 | 0 | 0
Not completed — QTc > 500 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- GTx-758 1000mg; GTx-758 2000mg: GTx-758/Experimental/ nonsteroidal selective ER alpha agonist
  GTx-758: comparison of different dosages of GTx-758 with leuprolide acetate for depot suspension
- Total: Total of all reporting groups
Arm/Group | GTx-758 1000mg | GTx-758 2000mg | Lupron Depot | Total
Number analyzed (Participants) | 53 | 55 | 51 | 159
Age, Continuous [Median (Full Range); unit: years] | 68 [44 to 78] | 68 [47 to 80] | 69 [50 to 79] | 68 [44 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 53 | 55 | 51 | 159
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 4 | 5 | 15
  Not Hispanic or Latino | 47 | 51 | 46 | 144
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 11 | 12 | 10 | 33
  White | 41 | 42 | 41 | 124
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 53 | 55 | 51 | 159

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Are Castrate by Day 60
Time Frame: 60 days
Population: Per-Protocol Population
Measure: Number; unit: participants
Groups:
- GTx- 758 1000mg; GTx-758 2000mg: GTx-758/Experimental/ nonsteroidal selective ER alpha agonist
  GTx-758: comparison of different dosages of GTx-758 with leuprolide acetate for depot suspension
Arm/Group | GTx- 758 1000mg | GTx-758 2000mg | Lupron Depot
Number analyzed (Participants) | 32 | 40 | 45
participants | 19 | 34 | 43

2. Secondary Outcome: Number of Participants Who Are Castrate by Day 60 and Maintained Castrate Range From Day 60 to Day 360/End of Study.
Time Frame: 12 months
Population: Castrate Population
Measure: Count of Participants; unit: Participants
Arm/Group | GTx- 758 1000mg | GTx-758 2000mg | Lupron Depot
Number analyzed (Participants) | 19 | 34 | 43
Participants | 0 | 3 | 9

3. Secondary Outcome: Time to Castration in Participants With Prostate Cancer
Description: Median time to castration was summarized using the Kaplan-Meier method.
Time Frame: 60 days
Population: Per-Protocol Population
Measure: Median (Full Range); unit: days
Arm/Group | GTx-758 1000mg | GTx-758 2000mg | Lupron Depot
Number analyzed (Participants) | 32 | 40 | 45
days | 29 [14 to 62] | 21 [7 to 68] | 21 [13 to 42]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | GTx- 758 1000mg | GTx-758 2000mg | Lupron Depot
All-Cause Mortality (participants affected / at risk) | 1/53 | 0/55 | 1/51
Serious Adverse Events (participants affected / at risk) | 11/53 | 6/55 | 4/51
Other Adverse Events (participants affected / at risk) | 46/53 | 49/55 | 48/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GTx- 758 1000mg (N=53) | GTx-758 2000mg (N=55) | Lupron Depot (N=51)
Acute Coronary Syndrome (Cardiac disorders) | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1
Atrial Fibrillation (Cardiac disorders) | 2 | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Cardiac Arrest (Cardiac disorders) | 1 | 0 | 0
Deep Vein Thrombosis (Vascular disorders) | 3 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0
Flank Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Hip Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 1 | 0
Hypnonatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Lung Infection (Infections and infestations) | 1 | 0 | 0
Metastases to Bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Myocardial Infarction (Cardiac disorders) | 1 | 0 | 0
Orthostatic Hypotension (Vascular disorders) | 0 | 0 | 1
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pathological Fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Sinus Bradycardia (Cardiac disorders) | 1 | 0 | 0
Urosepsis (Infections and infestations) | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GTx- 758 1000mg (N=53) | GTx-758 2000mg (N=55) | Lupron Depot (N=51)
anemia (Blood and lymphatic system disorders) | 1 | 3 | 0
lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 0
acute coronary syndrome (Cardiac disorders) | 4 | 0 | 0
angina (Cardiac disorders) | 0 | 1 | 0
right bundle branch block (Cardiac disorders) | 0 | 1 | 0
cardiac arrest (Cardiac disorders) | 1 | 0 | 0
conduction disorder (Cardiac disorders) | 0 | 1 | 0
coronary artery occlusion (Cardiac disorders) | 1 | 0 | 0
left ventricular dysfunction (Cardiac disorders) | 1 | 0 | 0
mitral valve disease (Cardiac disorders) | 1 | 0 | 0
myocardial infarction (Cardiac disorders) | 1 | 0 | 0
sinus bradycardia (Cardiac disorders) | 1 | 0 | 0
sinus tachycardia (Cardiac disorders) | 0 | 0 | 1
ventricular arrhythmia (Cardiac disorders) | 0 | 2 | 0
vertigo (Ear and labyrinth disorders) | 1 | 0 | 0
hypothyroidism (Endocrine disorders) | 0 | 1 | 0
conjunctival hemorrhage (Eye disorders) | 0 | 0 | 1
conjuntivitis (Eye disorders) | 0 | 1 | 0
visual acuity reduced (Eye disorders) | 0 | 0 | 1
vitreous floaters (Eye disorders) | 0 | 1 | 0
abdominal distension (Gastrointestinal disorders) | 1 | 1 | 0
abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0
abdominal pain, upper (Gastrointestinal disorders) | 0 | 2 | 0
colitis (Gastrointestinal disorders) | 0 | 2 | 0
colonic polyp (Gastrointestinal disorders) | 0 | 1 | 1
constipation (Gastrointestinal disorders) | 1 | 4 | 2
diarrhea (Gastrointestinal disorders) | 7 | 9 | 4
diverticulum (Gastrointestinal disorders) | 0 | 0 | 1
dry mouth (Gastrointestinal disorders) | 0 | 3 | 0
dyspepsia (Gastrointestinal disorders) | 6 | 5 | 1
gastritis (Gastrointestinal disorders) | 0 | 1 | 0
GI pain (Gastrointestinal disorders) | 0 | 1 | 0
gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 1 | 0
hemmorhoidal hemmorhage (Gastrointestinal disorders) | 1 | 0 | 0
hemorrhoids (Gastrointestinal disorders) | 0 | 1 | 1
impaired gastric emptying (Gastrointestinal disorders) | 0 | 1 | 0
large intestinal ulcer (Gastrointestinal disorders) | 1 | 0 | 0
lip swelling (Gastrointestinal disorders) | 0 | 2 | 0
nausea (Gastrointestinal disorders) | 7 | 3 | 4
oral pain (Gastrointestinal disorders) | 1 | 0 | 0
rectal discharge (Gastrointestinal disorders) | 1 | 0 | 0
swollen tongue (Gastrointestinal disorders) | 0 | 1 | 0
tooth ache (Gastrointestinal disorders) | 1 | 0 | 0
vomiting (Gastrointestinal disorders) | 3 | 3 | 0
chest pain (General disorders) | 0 | 0 | 1
chills (General disorders) | 0 | 1 | 2
fatigue (General disorders) | 6 | 8 | 9
influenza like illness (General disorders) | 0 | 4 | 4
infusion site pain (General disorders) | 1 | 0 | 0
injection site reaction (General disorders) | 1 | 0 | 2
irritability (General disorders) | 0 | 1 | 0
localized edema (General disorders) | 1 | 0 | 0
non cardiac chest pain (General disorders) | 2 | 1 | 1
edema, peripheral (General disorders) | 2 | 3 | 0
pyrexia (General disorders) | 4 | 2 | 0
vessel puncture site hematoma (General disorders) | 1 | 0 | 0
hepatobiliary disease (Hepatobiliary disorders) | 0 | 0 | 1
hypersensitivity (Immune system disorders) | 2 | 2 | 0
bronchitis (Infections and infestations) | 2 | 0 | 0
cellulitis (Infections and infestations) | 0 | 1 | 0
eye infection (Infections and infestations) | 0 | 1 | 0
gingival infection (Infections and infestations) | 0 | 0 | 1
laryngitis (Infections and infestations) | 0 | 1 | 0
lung infection (Infections and infestations) | 1 | 0 | 0
nail infection (Infections and infestations) | 0 | 0 | 1
nasopharyngitis (Infections and infestations) | 2 | 1 | 1
oral herpes (Infections and infestations) | 0 | 1 | 1
otitis externa (Infections and infestations) | 0 | 1 | 0
pharyngitis (Infections and infestations) | 0 | 1 | 2
pneumonia (Infections and infestations) | 1 | 0 | 0
sinusitis (Infections and infestations) | 0 | 0 | 2
skin infections (Infections and infestations) | 1 | 0 | 1
tooth infections (Infections and infestations) | 1 | 0 | 0
upper respiratory tract infections (Infections and infestations) | 3 | 0 | 1
urinary tract infections (Infections and infestations) | 4 | 5 | 3
urosepsis (Infections and infestations) | 0 | 1 | 0
contusion (Injury, poisoning and procedural complications) | 2 | 0 | 0
excoriation (Injury, poisoning and procedural complications) | 0 | 1 | 0
fall (Injury, poisoning and procedural complications) | 1 | 0 | 0
hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 0
radiation associated pain (Injury, poisoning and procedural complications) | 0 | 0 | 1
recall phenomenon (Injury, poisoning and procedural complications) | 1 | 0 | 0
rib fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
spinal column injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
alanine aminotransferase increase (Investigations) | 1 | 1 | 2
aspartate aminotransferase increase (Investigations) | 1 | 1 | 1
blood alkaline phosphatase increase (Investigations) | 0 | 1 | 0
blood bilirubin increase (Investigations) | 0 | 1 | 0
blood creatinine increase (Investigations) | 0 | 2 | 0
gamma-glutamyltransferase increase (Investigations) | 0 | 2 | 0
troponin-I increase (Investigations) | 0 | 1 | 0
weight decreased (Investigations) | 1 | 3 | 0
weight increased (Investigations) | 1 | 0 | 5
decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 1
dehydration (Investigations) | 0 | 1 | 0
hyperlipidemia (Metabolism and nutrition disorders) | 1 | 0 | 0
hypokalemia (Metabolism and nutrition disorders) | 1 | 0 | 0
hyponatremia (Metabolism and nutrition disorders) | 1 | 0 | 0
hypophosphatemia (Metabolism and nutrition disorders) | 1 | 0 | 0
increased appetite (Metabolism and nutrition disorders) | 0 | 0 | 2
iron overload (Metabolism and nutrition disorders) | 0 | 0 | 1
vitamin D deficiency (Metabolism and nutrition disorders) | 1 | 1 | 0
arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 4
arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2
back pain (Musculoskeletal and connective tissue disorders) | 1 | 3 | 5
exostosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
groin pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 4 | 0
musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1
neck mass (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
neck pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 2 | 1
pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
hepatic cancer, metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
seborrheic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
amnesia (Nervous system disorders) | 0 | 0 | 1
cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1
dizziness (Nervous system disorders) | 2 | 6 | 5
dysgeusia (Nervous system disorders) | 1 | 0 | 0
headache (Nervous system disorders) | 2 | 5 | 1
lethargy (Nervous system disorders) | 1 | 0 | 2
neuralgia (Nervous system disorders) | 1 | 0 | 0
paraesthesia (Nervous system disorders) | 3 | 0 | 1
parosmia (Nervous system disorders) | 0 | 1 | 0
radiculitis (Nervous system disorders) | 0 | 0 | 1
sinus headache (Nervous system disorders) | 0 | 0 | 1
somnolence (Nervous system disorders) | 1 | 0 | 0
syncope (Nervous system disorders) | 0 | 0 | 1
tremor (Nervous system disorders) | 1 | 0 | 0
anxiety (Psychiatric disorders) | 2 | 0 | 2
confusional state (Psychiatric disorders) | 0 | 1 | 0
depression (Psychiatric disorders) | 1 | 2 | 0
hallucination (Psychiatric disorders) | 0 | 1 | 0
insomnia (Psychiatric disorders) | 1 | 0 | 2
libido decreased (Psychiatric disorders) | 0 | 3 | 2
mood swings (Psychiatric disorders) | 0 | 0 | 1
azotemia (Renal and urinary disorders) | 0 | 1 | 0
bladder spasm (Renal and urinary disorders) | 0 | 1 | 0
calculus ureteric (Renal and urinary disorders) | 1 | 0 | 0
cystitis noninfective (Renal and urinary disorders) | 0 | 0 | 1
hematuria (Renal and urinary disorders) | 1 | 1 | 2
lower urinary tract symptoms (Renal and urinary disorders) | 0 | 1 | 0
micturition urgency (Renal and urinary disorders) | 0 | 2 | 1
nocturia (Renal and urinary disorders) | 1 | 0 | 1
pollakiuria (Renal and urinary disorders) | 2 | 6 | 4
renal failure (Renal and urinary disorders) | 1 | 1 | 0
renal pain (Renal and urinary disorders) | 0 | 1 | 0
terminal dribbling (Renal and urinary disorders) | 0 | 1 | 0
urinary hesitation (Renal and urinary disorders) | 0 | 1 | 0
urinary incontinence (Renal and urinary disorders) | 2 | 1 | 3
urinary retention (Renal and urinary disorders) | 0 | 1 | 0
urinary tract pain (Renal and urinary disorders) | 2 | 1 | 1
urinary flow decreased (Renal and urinary disorders) | 1 | 0 | 0
breast discharge (Reproductive system and breast disorders) | 1 | 0 | 0
breast discomfort (Reproductive system and breast disorders) | 0 | 1 | 0
breast pain (Reproductive system and breast disorders) | 15 | 21 | 0
breast tenderness (Reproductive system and breast disorders) | 1 | 4 | 0
ejaculation disorder (Reproductive system and breast disorders) | 0 | 1 | 0
erectile dysfunction (Reproductive system and breast disorders) | 0 | 1 | 1
gynecomastia (Reproductive system and breast disorders) | 5 | 4 | 1
nipple pain (Reproductive system and breast disorders) | 1 | 1 | 0
edema, genital (Reproductive system and breast disorders) | 1 | 1 | 0
pelvic pain (Reproductive system and breast disorders) | 0 | 1 | 0
perineal erythema (Reproductive system and breast disorders) | 0 | 1 | 0
prostatic obstruction (Reproductive system and breast disorders) | 0 | 2 | 0
testicular atrophy (Reproductive system and breast disorders) | 1 | 0 | 0
testicular pain (Reproductive system and breast disorders) | 1 | 1 | 0
asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
cough (Respiratory, thoracic and mediastinal disorders) | 1 | 5 | 0
dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 5 | 1
hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1
pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0
pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
rhinitis, allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0
upper airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
actinic keratosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
angioedema (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
dermatitis, allergic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
dermatitis, atopic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
dry skin (Skin and subcutaneous tissue disorders) | 0 | 3 | 0
erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
lentigo (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
onychoclasis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
pruritus (Skin and subcutaneous tissue disorders) | 2 | 0 | 2
rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
rash, maculo-papular (Skin and subcutaneous tissue disorders) | 3 | 3 | 0
skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
swelling face (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
urticaria (Skin and subcutaneous tissue disorders) | 1 | 2 | 0
deep vein thrombosis (Vascular disorders) | 8 | 2 | 0
hot flush (Vascular disorders) | 15 | 11 | 39
hypotension (Vascular disorders) | 0 | 1 | 0
lymphedema (Vascular disorders) | 0 | 0 | 1
orthostatic hypotension (Vascular disorders) | 0 | 0 | 1
thrombophlebitis (Vascular disorders) | 1 | 0 | 0
thrombophlebitis, superficial (Vascular disorders) | 1 | 1 | 0

LIMITATIONS AND CAVEATS:
Study terminated early

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No